CLINICAL TRIAL: NCT00215202
Title: A Phase II Trial of ZD1839 (Iressa) in Patients With Nonresectable Adrenocortical Carcinoma (ACC)
Brief Title: Phase II Trial of ZD1839 (Iressa) in Patients With Nonresectable Adrenocortical Carcinoma (ACC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: AstraZeneca (Industry); M.D. Anderson Cancer Center (Other); Dana-Farber Cancer Institute (Other); Kentuckiana Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: D0327
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Nonresectable Adrenocortical Carcinoma
Keywords: Adrenocortical Cancer; Iressa; Adrenal Cancer
MeSH Terms: conditions — Adrenal Cortex Neoplasms; Adrenal Gland Neoplasms | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Iressa (ZD1839)

SUMMARY:
The use of Iressa will result in a greater than 20% response rate in patients with nonresectable adrenocortical cancer who have previously been treated with one other form of systemic therapy (either Mitotane or chemotherapy).

DETAILED DESCRIPTION:
Adrenocortical carcinoma is a rare cancer with an incidence of 1.5 to 2 per million people in the United States. Surgery is the only potentially curative option. Current systemic therapy, either Mitotane or chemotherapy, typically gives response rates of 20% or less. This study is designed to see if the newer targeted therapy, Iressa, may be of benefit for patients with this fatal disease.

Patients with nonresectable adrenocortical cancer who have progressed on at least one other form of systemic therapy (Mitotane or chemotherapy) will be given Iressa 250 mg by mouth daily until disease progression. This is a standard two-stage Phase II clinical trial. Eighteen patients with measurable disease will be enrolled in the first stage. If there is at least one responder, then an additional nine patients with measurable disease will be enrolled for a total of 27 patients with measurable disease. Up to six patients without measurable disease may be enrolled at any point in this study. Iressa will be provided free for all study participants.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be able to provide informed consent
* Subject must be 18 years of age or older
* Subject must have histologically confirmed ACC by Department of Pathology at Dartmouth Hitchcock Medical Center
* Subject must have inoperable disease
* Subject must have received some form of systemic therapy prior to enrolling in the study

Exclusion Criteria:

* known severe hypersensitivity to Iressa
* other co-existing malignancies diagnosed within the last five years except basal cell cancer or cervical cancer in situ
* any unresolved CTC grade 2 toxicity from previous anticancer therapy (except alopecia)
* absolute neutrophil count less than 1.5 x 1,000,000,000 per liter
* platelets less than 20 x 1,000,000,000 per liter
* severe uncontrolled systemic disease
* pregnancy\breastfeeding
* women who are fertile and not willing to practice abstinence or contraception
* use of phenytoin, carbamazepine, rifampicin, barbiturates, or St. John's Wort
* treatment with a non-approved or investigational drug within 28 days before Day 1 of study treatment
* prior use of ZD1839 (Iressa) or any other anti-EGFR therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2004-08; Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to measure the objective response rate by RECIST (radiographic) criteria of nonresectable adrenocortical cancer to ZD1839

SECONDARY OUTCOMES:
Duration of response
Adverse event profile
Duration of survival
Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Samnotra, MD, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (4):
- United States (4):
  - Kentuckiana Cancer Institute PLLC, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - The University of Texas M.D. Anderson Cancer Center, Houston, Texas